CLINICAL TRIAL: NCT04055428
Title: The Effects of Natriuretic Peptide Augmentation on Cardiometabolic Health in Black Individuals (NAUTICAL)
Brief Title: NAUTICAL: Effect of Natriuretic Peptide Augmentation on Cardiometabolic Health in Black Individuals
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Associate Professor, Division of Cardiovascular Disease, Department of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 300003702; R01HL163852 (NIH)
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases; Insulin Sensitivity/Resistance; Metabolic Disease; Natriuretic Peptides; Metabolism; Energy Expenditure
Keywords: Natriuretic Peptides; Diabetes; Insulin Sensitivity; Energy Expenditure
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Insulin Resistance; Metabolic Diseases | interventions — sacubitril; Valsartan; Tablets; Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacubitril/Valsartan (Experimental): We will enroll 100 adult Black individuals. Each participant will take the assigned dose of medication twice daily for 12 weeks. We evaluate insulin sensitivity and energy expenditure at baseline and after 12 weeks of intervention.
  Interventions: Drug: Sacubitril, Valsartan 97-103 mg Oral Tablet; Other: Intravenous Glucose Tolerance Test; Dietary Supplement: Standardized Meals; Other: Exercise capacity VO2 maximum determination
- Valsartan (Active Comparator): We will enroll 100 adult Black individuals. Each participant will take the assigned dose of medication twice daily for 12 weeks. We evaluate insulin sensitivity and energy expenditure at baseline and after 12 weeks of intervention.
  Interventions: Drug: Valsartan 160 mg; Other: Intravenous Glucose Tolerance Test; Dietary Supplement: Standardized Meals; Other: Exercise capacity VO2 maximum determination

INTERVENTIONS:
Drug: Sacubitril, Valsartan 97-103 mg Oral Tablet — The subject will be randomized, in a double-blind manner to sacubitril/valsartan 97/103 mg twice daily for a period of 12 weeks.
  Other Names: Sacubitril/Valsartan arm
  Arms: Sacubitril/Valsartan
Drug: Valsartan 160 mg — The subject will be randomized, in a double-blind manner to valsartan 160 mg twice daily for a period of 12 weeks.
  Other Names: Valsartan arm
  Arms: Valsartan
Other: Intravenous Glucose Tolerance Test — An assessment of the insulin sensitivity will be done using the IVGTT, at baseline and after 12 weeks of pharmacological interventions.
Dietary Supplement: Standardized Meals — Participants will consume the standardized study mixed meal for the assessment of postprandial GLP-1 response to the meal.
Other: Exercise capacity VO2 maximum determination — Each participant's maximal oxygen capacity will be determined using modified Bruce treadmill protocol.

SUMMARY:
Black individuals are more likely to have decreased insulin sensitivity which results in a high risk for the development of cardiometabolic disease. The reasons for this are incompletely understood. Natriuretic peptides (NPs) are hormones produced by the heart that play a role in regulating the metabolic health of an individual. Low circulating level of NPs is an important contributor to increased risk for diabetes. The NP levels are relatively lower among Black individuals thus affecting their metabolic health and putting them at a higher risk for diabetes. This study aims to test the hypothesis that by augmenting NP levels using sacubitril/valsartan, among Black Individuals one can improve their metabolic health (as measured by insulin sensitivity & energy expenditure) and help establish the role of NPs in the underlying mechanism behind increased risk for cardiometabolic disease in these population.

DETAILED DESCRIPTION:
Black individuals are more likely to have a reduced insulin sensitivity which results in a greater risk for diabetes. However, the reasons for their decreased insulin sensitivity are not clearly understood. Natriuretic peptides (NPs) are hormones produced by the heart that is known to have a wide range of favorable metabolic effects. Studies indicate that lower NP levels are associated with a decreased insulin sensitivity and this may be causally related to the development of diabetes.

Evidence suggests that Black individuals have low levels of NPs. Increased clearance of NPs by neprilysin, an NP degrading enzyme, contributes to the low levels of NP among Black individuals. Since NPs play an important role in the regulation of insulin sensitivity and energy expenditure, one can infer that relatively low NP levels are an important biological contributor to the high prevalence rates of cardiometabolic disease in African Americans.

Sacubitril/valsartan is an FDA-approved inhibitor of neprilysin that augment NP levels. NP augmentation using sacubitril/valsartan has been shown to improve insulin sensitivity and lipid metabolism in a small clinical trial among obese White individuals. It can be postulated that NP augmentation in populations with relatively low NP levels will help in improving their metabolic health. Improvement in the metabolic health following NP augmentation will also help us to outline the relationship between the NP system and the risk of cardiometabolic disease among Black individuals.

We hypothesize that NP augmentation among Black individuals will show an improvement in their metabolic health as measured by insulin sensitivity and energy expenditure. We hypothesize that African American individuals will show an improvement in their insulin sensitivity and their resting & exercise energy expenditure after treatment with sacubitril/valsartan versus valsartan alone.

Our study will have the following aims. The first aim is to assess the change in the insulin sensitivity after NP augmentation therapy (using sacubitril/valsartan) as compared with NP neutral therapy (using valsartan) among Black individuals. We will measure the change in insulin sensitivity (assessed using IVGTT) after 12 weeks of intervention. We will also assess the change in NP levels (a marker of NP augmentation) & cyclic guanylate monophosphate (cGMP) levels after intervention and evaluate their relationship with the change in insulin sensitivity.

The second aim of our study is to examine the change in the energy expenditure after sacubitril/valsartan as compared to valsartan alone among Black individuals. The individuals enrolled in the first aim will also be examined for the change in resting as well as exercise energy expenditure. This will be assessed using standardized protocol performed using the metabolic cart and an exercise treadmill, at baseline and after 12 weeks of either sacubitril/valsartan or valsartan alone.

The secondary aim of our study is to assess the GLP-1 response to meals after treatment with sacubitril/valsartan in Black individuals. We will evaluate the change in postprandial GLP-1 response to meals at baseline and after 12 weeks of either sacubitril/valsartan or valsartan alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults: Age more than or equal to 18 years of age
* Self-identified race/ethnicity as African-American or Black
* Blood pressure: 120-160/80-100 mmHg

Exclusion Criteria:

* Women who are pregnant or breastfeeding or who can become pregnant and not practicing an acceptable method of birth control during the study (including abstinence)
* Have any past or present history of cardiovascular diseases (stroke, myocardial infarction, heart failure, transient ischemic attack, angina, or cardiac arrhythmia)
* BP more than 160/100 mmHg
* BMI >45 kg/m2
* History of diabetes or fasting plasma glucose >=126 mg/dL or HbA1C>=6.5%
* History of angioedema
* Current or past (<12 months) history of smoking
* Estimated GFR < 60 ml/min/1.73 m2; albumin-creatinine ratio ≥30 mg/g
* Hepatic Transaminase (AST and ALT) levels >3x the upper limit of normal
* Significant psychiatric illness or seizure disorder
* More than 2 Alcoholic drinks daily
* Anemia (men, Hct < 38%, Hb<13 g/dL; women, Hct <36%, Hb <12 g/dL)
* Inability to exercise on a treadmill

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity after natriuretic peptide augmentation | 12 weeks
  An assessment of the insulin sensitivity will be done at baseline and after 12 weeks of pharmacological intervention.
Change in energy expenditure after natriuretic peptide augmentation | 12 weeks
  An assessment of the resting energy expenditure will be done at baseline and after 12 weeks of pharmacological intervention.

SECONDARY OUTCOMES:
Change in exercise energy expenditure after 12 weeks of pharmacological intervention. | 12 weeks
  During standardized protocol after 12 weeks of intervention, the energy expenditure will be calculated using metabolic cart.
Change in post-meal increase in GLP-1 levels | 12 weeks
  Change in GLP-1 levels after a standardized meal after 12 weeks of pharmacological intervention
Change in peak oxygen consumption after 12 weeks of pharmacological intervention. | 12 weeks
  Change in the peak oxygen consumption (VO2 max) after 12 weeks of intervention.
Change in fasting GLP-1 levels | 12 weeks
  Change in fasting GLP-1 levels after 12 weeks of pharmacological intervention
Change in natriuretic peptide levels | 12 weeks
  Change in natriuretic peptide levels (ANP, MRproANP, BNP, NTproBNP) after 12 weeks of pharmacological intervention
Change in measures of insulin sensitivity | 12 weeks
  Change in measures of insulin sensitivity (AIRg, Sg, Kg, Disposition Index) after 12 weeks of pharmacological intervention
Change in HBA1c levels | 12 weeks
  Change in HBA1c levels after 12 weeks of pharmacological intervention
Change in fasting blood glucose levels | 12 weeks
  Change in fasting blood glucose levels after 12 weeks of pharmacological intervention
Change in HOMA-IR | 12 weeks
  Change in HOMA-IR after 12 weeks of pharmacological intervention
Change in fasting insulin levels | 12 weeks
  Change in fasting insulin levels after 12 weeks of pharmacological intervention
Change in measures of body mass index | 12 weeks
  Change in the measures of body mass index after 12 weeks of pharmacological intervention
Change in measures of hip circumference | 12 weeks
  Change in the measures of hip circumference after 12 weeks of pharmacological intervention
Change in measures of waist circumference | 12 weeks
  Change in the measures of waist circumference after 12 weeks of pharmacological intervention
Change in measures of adipose tissue mass | 12 weeks
  Change in the measures of adipose tissue mass after 12 weeks of pharmacological intervention
Change in total cholesterol levels | 12 weeks
  Change in the total cholesterol levels after 12 weeks of pharmacological intervention
Change in LDL-C levels | 12 weeks
  Change in LDL-C levels after 12 weeks of pharmacological intervention
Change in HDL-C levels | 12 weeks
  Change in HDL-C levels after 12 weeks of pharmacological intervention
Change in triglyceride levels | 12 weeks
  Change in triglyceride levels after 12 weeks of pharmacological intervention
Correlation of change in MR-pro atrial natriuretic peptide levels with change in insulin sensitivity after 12 weeks of pharmacological intervention. | 12 weeks
  The exposure-response relationship of change in MR-pro atrial natriuretic peptide levels with change in insulin sensitivity after 12 weeks of intervention will be examined.
Correlation of change in MR-pro atrial natriuretic peptide levels with change in energy expenditure after 12 weeks of pharmacological intervention. | 12 weeks
  The exposure-response relationship of change in MR-pro atrial natriuretic peptide levels with change in resting and exercise energy expenditure after 12 weeks of intervention will be examined.
Correlation of change in B-type natriuretic peptide levels with change in insulin sensitivity after 12 weeks of pharmacological intervention. | 12 weeks
  The exposure-response relationship of change in B-type natriuretic peptide levels with change in insulin sensitivity after 12 weeks of intervention will be examined.
Correlation of change in B-type natriuretic peptide levels with change in resting energy expenditure after 12 weeks of pharmacological intervention. | 12 weeks
  The exposure-response relationship of change in B-type natriuretic peptide levels with change in resting energy expenditure after 12 weeks of intervention will be examined.
Correlation of change in NT-pro B-type natriuretic peptide levels with change in insulin sensitivity after 12 weeks of pharmacological intervention. | 12 weeks
  The exposure-response relationship of change in NT-pro B-type natriuretic peptide levels with change in insulin sensitivity after 12 weeks of intervention will be examined.
Correlation of change in NT-pro B-type natriuretic peptide levels with change in energy expenditure after 12 weeks of pharmacological intervention. | 12 weeks
  The exposure-response relationship of change in NT-pro B-type natriuretic peptide levels with change in resting and exercise energy expenditure after 12 weeks of intervention will be examined.
Impact of Natriuretic Peptide Genotype on Study Endpoints | 12 weeks
  All study outcomes will be analyzed by natriuretic peptide genotypes

OTHER OUTCOMES:
Change in Metabolomic Profile | 12 weeks
  The change in the metabolomic profile examined using standardized platforms after 12 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, FAHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jordan J, Stinkens R, Jax T, Engeli S, Blaak EE, May M, Havekes B, Schindler C, Albrecht D, Pal P, Heise T, Goossens GH, Langenickel TH. Improved Insulin Sensitivity With Angiotensin Receptor Neprilysin Inhibition in Individuals With Obesity and Hypertension. Clin Pharmacol Ther. 2017 Feb;101(2):254-263. doi: 10.1002/cpt.455. Epub 2016 Nov 17. PMID 27542885
- [Result] Arora P, Reingold J, Baggish A, Guanaga DP, Wu C, Ghorbani A, Song Y, Chen-Tournaux A, Khan AM, Tainsh LT, Buys ES, Williams JS, Heublein DM, Burnett JC, Semigran MJ, Bloch KD, Scherrer-Crosbie M, Newton-Cheh C, Kaplan LM, Wang TJ. Weight loss, saline loading, and the natriuretic peptide system. J Am Heart Assoc. 2015 Jan 16;4(1):e001265. doi: 10.1161/JAHA.114.001265. PMID 25595796
- [Result] Seferovic JP, Claggett B, Seidelmann SB, Seely EW, Packer M, Zile MR, Rouleau JL, Swedberg K, Lefkowitz M, Shi VC, Desai AS, McMurray JJV, Solomon SD. Effect of sacubitril/valsartan versus enalapril on glycaemic control in patients with heart failure and diabetes: a post-hoc analysis from the PARADIGM-HF trial. Lancet Diabetes Endocrinol. 2017 May;5(5):333-340. doi: 10.1016/S2213-8587(17)30087-6. Epub 2017 Mar 18. PMID 28330649
- [Result] Patel N, Cushman M, Gutierrez OM, Howard G, Safford MM, Muntner P, Durant RW, Prabhu SD, Arora G, Levitan EB, Arora P. Racial differences in the association of NT-proBNP with risk of incident heart failure in REGARDS. JCI Insight. 2019 Jun 4;5(13):e129979. doi: 10.1172/jci.insight.129979. PMID 31162140